CLINICAL TRIAL: NCT05851313
Title: Role of Anthropometric Indices and Vit-D Supplementation on BioNTech, Pfizer Vaccine Side Effect and Immunoglobulin G Response Against SARS-CoV-2 in Individuals Infected With COVID-19; A Randomized Control Trial
Brief Title: Role of Vit-D Supplementation on BioNTech, Pfizer Vaccine Side Effect and Immunoglobulin G Response
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sulaimany Polytechnic university (Other)
Responsible Party: Principal Investigator, Hawal Lateef Fateh, Dr Hawal Lateef Fateh, Sulaimany Polytechnic university
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: KTC20230105
Record Dates: First submitted 2023-05-05; First posted 2023-05-09 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Respiratory Infection
Keywords: Vitamin D, Immunoglobulin G, COVID-19 vaccine, Side effects
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vitamin D supplementation for 16 weeks (Experimental): The intervention group received 600IU of vitamin D supplements every day, one hour after breakfast for 14-16 weeks.
  Interventions: Combination Product: Vitamin-D
- Placebo (Placebo Comparator): The control group took a placebo prepared with the same shape and size of supplements.
  Interventions: Combination Product: Vitamin-D

INTERVENTIONS:
Combination Product: Vitamin-D — The intervention group received 600IU of vitamin D supplements every day, one hour after breakfast for 14-16 weeks.

SUMMARY:
The goal of this clinical trial study is to investigate the role of anthropometric indices and Vit-D supplementation on BioNTech, Pfizer vaccine side effect and immunoglobulin G response against SARS-CoV-2 in individuals infected with COVID-19.

The main question[s] it aims to answer are:

1. BMI has role in reduce BioNTech, Pfizer vaccine side effect
2. BMI has role in improve IgG titer
3. Vit-D supplementation has role in reduce BioNTech, Pfizer vaccine side effect
4. Vit-D supplementation has role in improve IgG titer

DETAILED DESCRIPTION:
The intervention group received 600IU of vitamin D supplements every day, one hour after breakfast, for 14-16 weeks. The control group took a placebo prepared with the same shape and size of supplements. The supplement was given to the patients by someone other than the researcher, to ensure that the researchers did not know which group receiving the supplement/placebo (given the double-blindness of the study). Also, in this study, the person who did the data analysis did not aware of randomization. at first, a 3-day recall food questionnaire was taken from two groups. From the day, the subjects tested positive, they were asked to start supplementation for 4 weeks and return after that to take the first dose of the vaccine. Subjects were asked to continue to use supplements after the first vaccination. After 6 to 8 weeks, patients came back for another vaccination dose and were again asked to use the supplement for 4 weeks again, after that subjects were asked to come for a blood test.

ELIGIBILITY:
Inclusion criteria:

participants with COVID-19 positive tests.

Exclusion criteria:

1. Who did not take the vaccine
2. who take one dose of the vaccine
3. who did not come back for another dose
4. subjects who in the last 6 months received vitamin or mineral supplementation
5. those with chronic conditions such as diabetes, hypertension, and heart disease, unwillingness to continue the study protocol, lactating women and pregnant women.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Vit-D supplementation has role in reduce BioNTech, Pfizer vaccine side effect | 16 weeks
  Vitamin D supplement was given for 16 weeks

SECONDARY OUTCOMES:
Vit-D supplementation has role in improve IgG titer | 16 weeks
  Vitamin D supplement was given for 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hawal F Lateef, Msc, Principal Investigator — 1- Nursing Department, Kalar Technical College, Sulaimani polytechnic university, Sulaimani, Iraq
Locations (1):
- Hawal Lateef Fateh, Sulaymaniyah, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fateh HL, Kareem G, Rezaeian S, Moludi J, Kamari N. The Effect of Vit-D Supplementation on the Side Effect of BioNTech, Pfizer Vaccination and Immunoglobulin G Response Against SARS-CoV-2 in the Individuals Tested Positive for COVID-19: A Randomized Control Trial. Clin Nutr Res. 2023 Oct 24;12(4):269-282. doi: 10.7762/cnr.2023.12.4.269. eCollection 2023 Oct. PMID 37969936